CLINICAL TRIAL: NCT00657254
Title: Extension Program for Bay 43-9006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10922
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Neoplasm; Metastasis
Keywords: Extension; Sorafenib; Survival
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Bay 43-9006 400mg (2 x 200mg tablets) orally twice daily until withdrawal.

SUMMARY:
The study was designed to allow for the continuation of treatment with Sorafenib as a single agent to those patients who participated in a previous Sorafenib study that had reached its designated end-date and who were, in the opinion of the Investigator and the Sponsor, still benefiting from treatment.

ELIGIBILITY:
Inclusion Criteria: - Patients who had participated in a previous sorafenib study that had completed, who did not meet withdrawal criteria of the previous study and who were, in the opinion of the investigator and sponsor still benefiting from treatment. Exclusion Criteria:- The current cardiovascular situation of the patient was carefully re-evaluated by both the investigator and the sponsor and an informed decision as to inclusion was then made.- Substance abuse, medical, psychological or social conditions that may have interfered with the patient's participation in the study or evaluation of the study results.- Known or suspected allergy to the investigational agent.- Any condition that was unstable or which could jeopardise the safety of the patient and his/her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Survival | Death

SECONDARY OUTCOMES:
Objective Tumour Response Rate | Number of confirmed partial and complete responses
Overall Response Duration | Time from the date of the first intake of sorafenib to the date that progressive disease is documented.
Time to Objective Response | Time from the date of the first intake of sorafenib to the date that objective response is first documented.
Time to Disease Progression | Time from first intake of sorafenib to disease progression
Safety Parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Boston, Massachusetts, United States
- Bruxelles - Brussel, Belgium
- Canada (2):
  - Hamilton, Ontario
  - Toronto, Ontario
- Germany (2):
  - Essen, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia